CLINICAL TRIAL: NCT02567435
Title: A Randomized Phase 3 Study of Vincristine, Dactinomycin, Cyclophosphamide (VAC) Alternating With Vincristine and Irinotecan (VI) Versus VAC/VI Plus Temsirolimus (TORI, Torisel, NSC# 683864) in Patients With Intermediate Risk (IR) Rhabdomyosarcoma (RMS)
Brief Title: Combination Chemotherapy With or Without Temsirolimus in Treating Patients With Intermediate Risk Rhabdomyosarcoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01644; NCI-2015-01644 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARST1431; ARST1431 (Other: Children's Oncology Group); ARST1431 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Alveolar Rhabdomyosarcoma; Botryoid-Type Embryonal Rhabdomyosarcoma; Embryonal Rhabdomyosarcoma; Rhabdomyosarcoma; Sclerosing Rhabdomyosarcoma; Spindle Cell Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma, Alveolar; Rhabdomyosarcoma, Embryonal; Rhabdomyosarcoma | interventions — Cyclophosphamide; Dactinomycin; Irinotecan; Radiotherapy; Radiation; temsirolimus; Sirolimus; Vincristine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen A (VAC/VI) (Experimental): Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1-13, 16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, cyclophosphamide IV over 60 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 4, 10, 16, 19, 25, 31, and 37. Patients also undergo primary site RT beginning at week 13 or metastatic site RT beginning at week 43 for up to 6.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients then receive vinorelbine IV over 6-10 minutes on days 1, 8, and 15 and cyclophosphamide PO QD on days 1-28. Cycles repeats every 28 days for 24 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Regimen B (VAC/VI/temsirolimus) (Experimental): Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1-13, 16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, cyclophosphamide IV over 60 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 4, 10, 16, 19, 25, 31, and 37 and temsirolimus IV over 30-60 minutes on day 1 of weeks 1-12 and 21-42. Patients also undergo RT as in Regimen A. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients then receive vinorelbine IV over 6-10 minutes on days 1, 8, and 15 and cyclophosphamide PO QD on days 1-28. Cycles repeats every 28 days for 24 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Temsirolimus; Drug: Vincristine Sulfate; Drug: Vinorelbine
- Regimen C (FOXO1 fusion negative, VAC/VA) (Experimental): Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1-10 and 13-22, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of weeks 1, 4, 7, 10, 13, 16, 19, and 22, cyclophosphamide IV over 60 minutes on day 1 of weeks 1, 4, 7, and 10. Patients undergo RT beginning at week 13 for up to 6.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Biological: Dactinomycin; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV and PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
  Arms: Regimen A (VAC/VI); Regimen B (VAC/VI/temsirolimus)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Temsirolimus — Given IV
  Other Names: CCI 779; CCI-779; CCI-779 Rapamycin Analog; CCI779; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
  Arms: Regimen B (VAC/VI/temsirolimus)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
Drug: Vinorelbine — Given IV
  Other Names: Dihydroxydeoxynorvinkaleukoblastine
  Arms: Regimen B (VAC/VI/temsirolimus)

SUMMARY:
This randomized phase III trial studies how well combination chemotherapy (vincristine sulfate, dactinomycin, cyclophosphamide alternated with vincristine sulfate and irinotecan hydrochloride or vinorelbine) works compared to combination chemotherapy plus temsirolimus in treating patients with rhabdomyosarcoma (cancer that forms in the soft tissues, such as muscle), and has an intermediate chance of coming back after treatment (intermediate risk). Drugs used work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Combination chemotherapy and temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether chemotherapy plus temsirolimus is more effective than chemotherapy alone in treating patients with intermediate-risk rhabdomyosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the event-free survival (EFS) of patients with intermediate-risk (IR) rhabdomyosarcoma (RMS) treated with surgery, radiotherapy, and vincristine (vincristine sulfate), dactinomycin, and cyclophosphamide (VAC) alternating with vincristine and irinotecan (irinotecan hydrochloride) (VI) (VAC/VI) with maintenance to that of patients treated with surgery, radiotherapy and VAC/VI plus temsirolimus with maintenance.

SECONDARY OBJECTIVE:

I. To compare the overall survival (OS) of patients with IR RMS treated with surgery, radiotherapy, and VAC alternating with VI with maintenance to that of patients treated with surgery, radiotherapy and VAC/VI plus temsirolimus with maintenance.

EXPLORATORY OBJECTIVES:

I. To compare the outcome of patients based on their FOXO1 fusion gene partner, by evaluating PAX3 versus (vs) PAX7 in all patients found to be FOXO1 fusion positive.

II. To compare the outcome of patients based on their [F18]-fluorodeoxy-D-glucose-positron emission tomography (FDG-PET) response at week 9 (positive or negative), as assessed by Deauville criteria (5-point).

III. To estimate the frequency of patients with circulating tumor deoxyribonucleic acid (DNA) (ctDNA) at diagnosis and subsequent time-points, and explore whether tumor-specific somatic variants are detectable in the ctDNA.

IV. To compare the outcome of patients (VAC/VI with or without temsirolimus) who have received maintenance therapy on ARST1431 to those who received VAC/VI on ARST0531.

OUTLINE:

FEASIBILITY PHASE (THE FEASIBILITY PHASE IS COMPLETE, EFFECTIVE WITH AMENDMENT #1A): (< 21 years old): This is a dose-escalation study of temsirolimus.

Patients receive vincristine sulfate intravenously (IV) over 1 minute on day 1 of weeks 1-13, 16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, cyclophosphamide IV over 60 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 4, 10, 16, 19, 25, 31, and 37, and temsirolimus IV over 30-60 minutes on days 1, 8, and 15. Patients also undergo radiation therapy (RT) beginning week 13 for up to 6.5 weeks. Courses with temsirolimus repeat every 21 days for 12 weeks in the absence of disease progression or unacceptable toxicity.

EFFICACY PHASE: Patients are randomized to Regimen A or B. Patients with disease that is ARMS FOXO1 fusion negative (stage I, group I/II, stage 1, group III [orbit] or stage II, group I/II) are assigned to Regimen C.

REGIMEN A (VAC/VI): Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1-13, 16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, cyclophosphamide IV over 60 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 4, 10, 16, 19, 25, 31, and 37. Patients also undergo primary site RT beginning at week 13 or metastatic site RT beginning at week 43 for up to 6.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients then receive vinorelbine IV over 6-10 minutes on days 1, 8, and 15 and cyclophosphamide orally (PO) once daily (QD) on days 1-28. Cycles repeats every 28 days for 24 weeks in the absence of disease progression or unacceptable toxicity.

REGIMEN B (VAC/VI TEMSIROLIMUS): Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1-13, 16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, cyclophosphamide IV over 60 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 4, 10, 16, 19, 25, 31, and 37 and temsirolimus IV over 30-60 minutes on day 1 of weeks 1-12 and 21-42. Patients also undergo RT as in Regimen A. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients then receive vinorelbine IV over 6-10 minutes on days 1, 8, and 15 and cyclophosphamide PO QD on days 1-28. Cycles repeats every 28 days for 24 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE (Patients in Regimen A or Regimen B): Patients receive vinorelbine IV over 6-10 minutes on days 1, 8, and 15 and cyclophosphamide orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 6 cycles.

REGIMEN C (FOXO1 FUSION NEGATIVE): Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1-10 and 13-22, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of weeks 1, 4, 7, 10, 13, 16, 19, and 22, cyclophosphamide IV over 60 minutes on day 1 of weeks 1, 4, 7, and 10. Patients undergo RT beginning at week 13 for up to 6.5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 2 years, every 6 months for 1 year, and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Feasibility Phase: Patients must be < 21 years of age at the time of enrollment; please note: the feasibility phase is complete, effective with amendment #1
* Efficacy Phase: Patients must be =< 40 years of age at the time of enrollment
* Patients with newly diagnosed RMS of any subtype, except adult-type pleomorphic, based upon institutional histopathologic classification, are eligible to enroll on the study based upon stage, group, and age, as below
* RMS types included under embryonal rhabdomyosarcoma (ERMS) include those classified in the 1995 International Classification of Rhabdomyosarcoma (ICR) as ERMS (classic, spindle cell, and botryoid variants), which are reclassified in the 2013 World Health Organization (WHO) classification as ERMS (classic, dense and botryoid variants) and spindle cell/sclerosing RMS (encompassing the historical spindle cell ERMS variant and the newly recognized sclerosing RMS variant); classification of alveolar rhabdomyosarcoma (ARMS) in the 2013 WHO classification is the same as in the ICR and includes classic and solid variants

  * ERMS

    * Stage 1, group III (non-orbit)
    * Stage 3, group I/II
    * Stage 2/3, group III
    * Stage 4, group IV, < 10 years old
  * ARMS:

    * Stages 1-3, groups I-III
* Specimen Submission: Patients must have sufficient tissue available for the required biology study
* Lansky performance status score >= 50 for patients =< 16 years of age; Karnofsky performance status score >= 50 for patients > 16 years of age
* Peripheral absolute neutrophil count (ANC) >= 750/uL
* Platelet count >= 75,000/uL
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 month to < 6 months old: 0.4 mg/dl (male), 0.4 mg/dl (female)
  * 6 months to < 1 year old: 0.5 mg/dl (male), 0.5 mg/dl (female)
  * 1 to < 2 years old: 0.6 mg/dl (male), 0.6 mg/dl (female)
  * 2 to < 6 years old: 0.8 mg/dl (male), 0.8 mg/dl (female)
  * 6 to < 10 years old: 1 mg/dl (male), 1 mg/dl (female)
  * 10 to < 13 years old: 1.2 mg/dl (male), 1.2 mg/dl (female)
  * 13 to < 16 years old: 1.5 mg/dl (male), 1.4 mg/dl (female)
  * >= 16 years old: 1.7 mg/dl (male), 1.4 mg/dl (female)
  * Patients with an elevated serum creatinine due to obstructive hydronephrosis secondary to tumor are still eligible; however, patients with urinary tract obstruction by tumor must have unimpeded urinary flow established via diversion (i.e. percutaneous nephrostomies or ureteric stents) of the urinary tract
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Patients who have previously received temsirolimus, another mTOR inhibitor, or any other investigational agent
* Patients who have received any chemotherapy (excluding steroids) and/or RT prior to this enrollment
* Patients with uncontrolled hyperglycemia
* Patients with uncontrolled hyperlipidemia
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for at least 3 months after treatment is completed
* Female patients who are pregnant are not eligible since fetal toxicities or teratogenic effects have been noted for several of the study drugs; Note: A pregnancy test is required for female patients of childbearing potential prior to study entry
* Lactating females who plan to breastfeed their infants are not eligible

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 325 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2026-10-27 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Abha A Gupta, Principal Investigator — Children's Oncology Group
Locations (384):
- United States (357):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Westchester Medical Center, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Carolina Surgical - Randolph, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (3):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Gupta AA, Xue W, Harrison DJ, Hawkins DS, Dasgupta R, Wolden S, Shulkin B, Qumseya A, Routh JC, MacDonald T, Feinberg S, Crompton B, Rudzinski ER, Arnold M, Venkatramani R. Addition of temsirolimus to chemotherapy in children, adolescents, and young adults with intermediate-risk rhabdomyosarcoma (ARST1431): a randomised, open-label, phase 3 trial from the Children's Oncology Group. Lancet Oncol. 2024 Jul;25(7):912-921. doi: 10.1016/S1470-2045(24)00255-9. PMID 38936378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was opened for enrollment on May 23, 2016, and was temporarily closed to accrual on September 23, 2016 for feasibility review. The study was re-opened for enrollment on January 2, 2018. The study was temporarily closed again on August 22, 2018 and re-opened on December 31, 2018 with the addition of maintenance therapy. The study is closed to accrual since 1/6/2022.
Pre-assignment Details: Among the 325 patients that enrolled, 4 patients were ineligible, 11 eligible patients were enrolled onto the feasibility phase (with 1 transferred to Regimen C), and 310 eligible patients were randomized and enrolled onto the efficacy phase (with 2 transferred to Regimen C). 13 randomized eligible patients were not analyzed (not evaluable due to FOXO1 diagnosis or amendment after study activated).
Groups:
- Feasibility (VAC/VI/Temsirolimus): Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1-13, 16, 17, 19, 20, 22-26, 28, 31-34, 37, 38, and 40, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, cyclophosphamide IV over 60 minutes on day 1 of weeks 1, 7, 13, 22, 28, 34, and 40, irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 4, 10, 16, 19, 25, 31, and 37 and temsirolimus IV over 30-60 minutes on day 1 of weeks 1-12 and 21-42. Patients also undergo RT as in Regimen A. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients then receive vinorelbine IV over 6-10 minutes on days 1, 8, and 15 and cyclophosphamide PO QD on days 1-28. Cycles repeats every 28 days for 24 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Regimen A (VAC/VI) | Regimen B (VAC/VI/Temsirolimus) | Regimen C (FOXO1 Fusion Negative, VAC/VA) | Feasibility (VAC/VI/Temsirolimus)
Started | 156 | 156 | 3 | 10
Completed | 150 | 147 | 3 | 9
Not Completed | 6 | 9 | 0 | 1
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Ineligible | 1 | 3 | 0 | 0
Not completed — Withdrawal of consent for any further data submissions | 4 | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A (VAC/VI) | Regimen B (VAC/VI/Temsirolimus) | Regimen C (FOXO1 Fusion Negative, VAC/VA) | Feasibility (VAC/VI/Temsirolimus) | Total
Number analyzed (Participants) | 156 | 156 | 3 | 10 | 325
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 145 | 140 | 3 | 10 | 298
  Between 18 and 65 years | 11 | 16 | 0 | 0 | 27
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 6.57 [0.04 to 35.84] | 6.05 [0.35 to 32.91] | 5.71 [3.18 to 6.58] | 4.59 [0.17 to 14.37] | 6.34 [0.04 to 35.84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 55 | 0 | 3 | 129
  Male | 85 | 101 | 3 | 7 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 17 | 2 | 1 | 49
  Not Hispanic or Latino | 113 | 117 | 1 | 9 | 240
  Unknown or Not Reported | 14 | 22 | 0 | 0 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 5 | 4 | 0 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 20 | 16 | 0 | 1 | 37
  White | 99 | 106 | 2 | 8 | 215
  More than one race | 3 | 3 | 0 | 1 | 7
  Unknown or Not Reported | 27 | 26 | 1 | 0 | 54
Region of Enrollment [Number; unit: participants]
  United States | 141 | 135 | 3 | 10 | 289
  Australia | 6 | 11 | 0 | 0 | 17
  Canada | 6 | 9 | 0 | 0 | 15
  New Zealand | 3 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: The Kaplan-Meier method will used to estimate 3-year EFS between the randomized treatment groups (Regimen A (VAC/VI) vs. Regimen B (VAC/VI/Temsirolimus)) using the log-rank test. EFS event is defined as the time from study entry until first occurrence of progression, relapse, second malignancy, or death.
Time Frame: Up to 3 years from study entry
Population: As pre-specified in the protocol, patients randomized to Regimen A (VAC/VI) and Regimen B (VAC/VI/Temsirolimus) were included in this analysis. The data was analyzed with revised intention-to-treat approach. Following patients were excluded 4 ineligible patients, 11 feasibility patients and 13 inevaluable patients (due to FOXO1 results or who did not receive maintenance therapy due to an amendment added during the study) .
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen A (VAC/VI) | Regimen B (VAC/VI/Temsirolimus)
Number analyzed (Participants) | 148 | 149
Percentage of participants | 64.80 [55.5 to 74.1] | 66.80 [57.5 to 76.2]
Statistical Analysis 1: Comparison: Regimen A (VAC/VI) vs Regimen B (VAC/VI/Temsirolimus); Test type: Superiority; p = 0.44, Log Rank; 3-Year EFS = 65.8

2. Secondary Outcome: Overall Survival (OS)
Description: The Kaplan-Meier method will used to estimate 3-year OS between the randomized treatment groups (Regimen A (VAC/VI) vs. Regimen B (VAC/VI/Temsirolimus)) using the log-rank test. OS event is defined as the time from study entry until death.
Time Frame: Up to 3 years from study entry
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen A (VAC/VI) | Regimen B (VAC/VI/Temsirolimus)
Number analyzed (Participants) | 148 | 149
Percentage of participants | 78.70 [70.9 to 86.4] | 77.80 [69.7 to 85.9]
Statistical Analysis 1: Comparison: Regimen A (VAC/VI) vs Regimen B (VAC/VI/Temsirolimus); Test type: Superiority; p = 0.56, Log Rank; 3-Year OS = 78.2

3. Other Pre Specified Outcome: Frequency of Circulating Tumor DNA (ctDNA) at Diagnosis and Subsequent Time-points
Description: Will determine the frequency with which of ctDNA is detected in patients with intermediate-risk (IR) rhabdomyosarcoma (RMS) at diagnosis and how these levels change over time with. In addition, the level of ctDNA as a percent of total cell-free DNA will be summarized by reporting the median and range. Since no prior data are available on the rate of positivity nor the change over time, the analysis will be purely descriptive. Changes over time will be plotted to visually determine and compare the trajectories of ctDNA during the early and late stages of therapy.
Time Frame: Up to 10 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Patient Outcome Based on Their Forkhead Box O1 Protein (FOXO1) Partner, by Evaluating PAX3 vs. PAX7 in All Patients Found to be FOXO1 Fusion Positive
Time Frame: Up to 10 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Patient Outcome Based on Their [F18]-Fluorodeoxy-D-glucose-positron Emission Tomography (FDG-positron Emission Tomography [PET]) Response
Description: Assessed by Deauville Criteria (5-point).
Time Frame: At week 9
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Patient Outcomes Based on (Vincristine, Dactinomycin, and Cyclophosphamide [VAC]/Vincristine and Irinotecan [VI] With or Without Temsirolimus) Who Have Received Maintenance Therapy on ARST1431 to Those Who Received VAC/VI on ARST0531
Description: The two-sample log-rank test will be performed.
Time Frame: Up to 10 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events monitored/assessed up to 66 weeks from study entry. All-Cause Mortality monitored/assessed up to 7 years and 4 months from study entry.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Regimen A (VAC/VI) | Regimen B (VAC/VI/Temsirolimus) | Regimen C (FOXO1 Fusion Negative, VAC/VA) | Feasibility (VAC/VI/Temsirolimus)
All-Cause Mortality (participants affected / at risk) | 33/155 | 33/153 | 0/3 | 4/10
Serious Adverse Events (participants affected / at risk) | 17/155 | 77/153 | 0/3 | 6/10
Other Adverse Events (participants affected / at risk) | 139/155 | 141/153 | 1/3 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (VAC/VI) (N=155) | Regimen B (VAC/VI/Temsirolimus) (N=153) | Regimen C (FOXO1 Fusion Negative, VAC/VA) (N=3) | Feasibility (VAC/VI/Temsirolimus) (N=10)
Abdominal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 6 (7) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cecal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 13 (16) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 7 (8) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 6 (9) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 8 (11) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 35 (44) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (9) | 8 (11) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (VAC/VI) (N=155) | Regimen B (VAC/VI/Temsirolimus) (N=153) | Regimen C (FOXO1 Fusion Negative, VAC/VA) (N=3) | Feasibility (VAC/VI/Temsirolimus) (N=10)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 2 (3) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 15 (23) | 29 (36) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 24 (31) | 39 (74) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 7 (7) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 14 (31) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 107 (417) | 117 (474) | 1 (2) | 3 (11)
Anorectal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 42 (68) | 42 (73) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (5) | 16 (17) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (11) | 17 (34) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 2 (3) | 4 (4) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (3)
Blood bilirubin increased (Investigations) | 3 (9) | 4 (4) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 5 (7) | 1 (1) | 0 (0) | 1 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (6) | 6 (6) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 24 (30) | 18 (23) | 0 (0) | 1 (1)
Corneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (5) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 26 (28) | 21 (25) | 0 (0) | 3 (3)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 17 (18) | 18 (19) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 43 (73) | 50 (78) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (5) | 0 (0) | 0 (0)
Edema face (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 11 (16) | 18 (24) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 12 (15) | 13 (18) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 56 (87) | 61 (92) | 0 (0) | 2 (4)
Fecal incontinence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 36 (52) | 46 (66) | 0 (0) | 1 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 4 (8) | 3 (4) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 6 (6) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 4 (5) | 3 (3) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 10 (31) | 12 (30) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 21 (34) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (23) | 27 (38) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 14 (17) | 22 (27) | 0 (0) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 21 (25) | 30 (44) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 7 (7) | 5 (5) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 15 (17) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 15 (21) | 16 (19) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 20 (23) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 9 (9) | 0 (0) | 1 (3)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 4 (4) | 6 (6) | 0 (0) | 1 (2)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 7 (7) | 7 (8) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 79 (316) | 81 (298) | 0 (0) | 2 (10)
Lymphocyte count increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 30 (35) | 55 (75) | 0 (0) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 56 (113) | 52 (88) | 0 (0) | 3 (3)
Neck edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 107 (506) | 109 (510) | 1 (3) | 6 (14)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 10 (12) | 5 (5) | 0 (0) | 1 (2)
Pain (General disorders) | 5 (6) | 8 (10) | 1 (1) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (11) | 10 (13) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papilledema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 16 (20) | 26 (36) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (30) | 26 (39) | 0 (0) | 2 (2)
Peritoneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phantom pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 49 (88) | 61 (115) | 0 (0) | 2 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 7 (8) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 8 (9) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 4 (6) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 8 (9) | 8 (10) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 9 (10) | 8 (8) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Social circumstances - Other, specify (Social circumstances) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tendon reflex decreased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (11) | 2 (2) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 8 (10) | 12 (13) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 18 (20) | 16 (24) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 5 (5) | 4 (7) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 12 (18) | 22 (31) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 3 (6) | 0 (0) | 2 (4)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urostomy stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 48 (98) | 46 (77) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 26 (42) | 31 (51) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 103 (454) | 103 (448) | 1 (1) | 4 (13)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 3 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT02567435/Prot_SAP_000.pdf